CLINICAL TRIAL: NCT02959827
Title: Iodinated Contrast Agents and Risk of Hypothyroidism in Young Children in the United States
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 19185
Record Dates: First submitted 2016-10-11; First posted 2016-11-09 (Estimated); Results first posted 2019-01-30 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Hypothyroidism
Keywords: Hypothyroidism,; children,; iodinated contrast agents,; retrospective cohort,; database
MeSH Terms: conditions — Hypothyroidism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Iodinated contrast agents: Children under age 4 in the Kaiser Permanente Northern California database, who had a diagnostic procedure with an iodinated contrast agent
  Interventions: Drug: Iodinated contrast agents

INTERVENTIONS:
Drug: Iodinated contrast agents — Use of iodine contrast agents and doses following the decision of the treating physician.

SUMMARY:
This study will estimate the incidence of hypothyroidism in a pediatric population of children under age 4, based on data from the US-based Kaiser Permanente Northern California database, which were exposed to iodinated contrast agent through having a diagnostic procedure.

ELIGIBILITY:
Inclusion Criteria:

* Children under age 4 in the Kaiser Permanente Northern California (KPNC) database, who had a diagnostic procedure with an iodinated contrast agent.
* Participants should be member of the KPNC for at least 3 months before the iodinated contrast exposure, except where the child is under 3 months of age at time of initial exposure, and 2 weeks after the exposure.

Exclusion Criteria:

* Diagnosis of hypothyroid any time prior to the iodine contrast exposure.
* Lab values for low thyroid (TSH > 5 mU/L for children) any time before the exposure
* Thyroid replacement therapy, Hashimoto thyroiditis, or congenital hypothyroidism any time prior to exposure.

Max Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children under age 4 in the Kaiser Permanente Northern California database, who had a diagnostic procedure with an iodinated contrast agent
Sampling Method: Non-Probability Sample
Enrollment: 2320 (Actual)
Dates: Start 2016-10-15 (Actual); Primary Completion 2017-06-15 (Actual); Study Completion 2017-06-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Oakland, Oakland, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was a retrospective cohort study, using the data from the years 2008 to June of 2016 in the database of Kaiser Permanente Northern California.
Pre-assignment Details: There were 2320 children identified in Kaiser Permanente Northern California who met our study population criteria: patients who had a procedure that used iodinated contrast agent and were under the age of 4, during the years 2008 to June of 2016.
Groups:
- Iodine Contrast Agent: Children under age 4, from the US-based Kaiser Permanente Northern California database, who were exposed to iodinated contrast agent through having a diagnostic procedure.
Period: Overall Study
Arm/Group | Iodine Contrast Agent
Started | 2320
Completed | 2320
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Iodine Contrast Agent
Number analyzed (Participants) | 2320
Age, Customized [Count of Participants; unit: Participants]
  <1 month | 197
  1 to 3 months | 174
  3 to 6 months | 174
  6 months to 1 year | 257
  1 to 4 years | 1518
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1032
  Male | 1288
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 800
  African American | 174
  Hispanic | 726
  Asian/Pacific islander | 425
  Other or missing | 195

OUTCOME MEASURES:

1. Primary Outcome: Incidence Rate of Hypothyroidism Detected in Routine Clinical Practice
Description: Incidence density rates (IDR) were calculated as the number of cases over the person time at risk where the numerator was the number of cases and the denominator was the person years at risk.
Time Frame: In the 365 days post exposure to an iodinated contrast agent
Measure: Mean (95% Confidence Interval); unit: events per 1,000 person years
Arm/Group | Iodine Contrast Agent
Number analyzed (Participants) | 2320
events per 1,000 person years | 15.9 [11.2 to 22.0]

2. Secondary Outcome: Baseline Characteristics (Age) of the Cases With Hypothyroidism and of the Rest of the Cohort
Time Frame: Up to 365 days after a diagnostic scan with iodinated contrast agent
Measure: Count of Participants; unit: Participants
Groups:
- Hypothyroidism Cases: Participants who met the criteria to be a case of hypothyroidism were identified.
- Non-hypothyroidism Cases: Participants who did not meet the criteria to be a case of hypothyroidism were identified.
Arm/Group | Hypothyroidism Cases | Non-hypothyroidism Cases
Number analyzed (Participants) | 34 | 2286
Participants
  <1 month | 4 | 193
  1 to 3 months | 6 | 168
  3 to 6 months | 6 | 168
  6 months to 1 year | 4 | 253
  1 to 4 years | 14 | 1504

3. Secondary Outcome: Baseline Characteristics (Sex) of the Cases With Hypothyroidism and of the Rest of the Cohort
Time Frame: Up to 365 days after a diagnostic scan with iodinated contrast agent
Measure: Count of Participants; unit: Participants
Arm/Group | Hypothyroidism Cases | Non-hypothyroidism Cases
Number analyzed (Participants) | 34 | 2286
Participants
  Male | 24 | 1264
  Female | 10 | 1022

4. Secondary Outcome: Baseline Characteristics (Year of Hypothyroidism Diagnosis) of the Cases With Hypothyroidism and of the Rest of the Cohort
Time Frame: Up to 365 days after a diagnostic scan with iodinated contrast agent
Measure: Count of Participants; unit: Participants
Arm/Group | Hypothyroidism Cases | Non-hypothyroidism Cases
Number analyzed (Participants) | 34 | 2286
Participants
  2008 | 4 | 300
  2009 | 3 | 320
  2010 | 9 | 297
  2011 | 2 | 260
  2012 | 2 | 266
  2013 | 4 | 263
  2014 | 4 | 234
  2015 | 6 | 241
  through August 2016 | 0 | 105

5. Secondary Outcome: Baseline Characteristics (Type of Iodine Contrast Exposure) of the Cases With Hypothyroidism and of the Rest of the Cohort
Time Frame: Up to 365 days after a diagnostic scan with iodinated contrast agent
Measure: Count of Units; unit: Iodine contrast exposure
Units Other Than Participants: Iodine contrast exposure
Arm/Group | Hypothyroidism Cases | Non-hypothyroidism Cases
Number analyzed (Participants) | 34 | 2286
Number analyzed (Iodine contrast exposure) | 34 | 2290
Iodine contrast exposure
  CT scan | 18 | 1762
  Heart catheterization | 16 | 528

6. Secondary Outcome: Baseline Characteristics (Race/Ethnicity) of the Cases With Hypothyroidism and of the Rest of the Cohort
Time Frame: Up to 365 days after a diagnostic scan with iodinated contrast agent
Measure: Count of Participants; unit: Participants
Arm/Group | Hypothyroidism Cases | Non-hypothyroidism Cases
Number analyzed (Participants) | 34 | 2286
Participants
  White | 13 | 787
  African American | 4 | 170
  Hispanic | 6 | 720
  Asian/Pacific islander | 9 | 416
  Other or missing | 2 | 193

7. Secondary Outcome: Time From First Iodinated Contrast to First Hypothyroidism Event
Time Frame: Up to 365 days after a diagnostic scan with iodinated contrast agent
Measure: Count of Participants; unit: Participants
Groups:
- Hypothyroidism Cases With CT Scan: Participants who had CT scan and met the criteria to be a case of hypothyroidism were identified.
- Hypothyroidism Cases With Cardiac Catheterization: Participants who had cardiac catheterization and met the criteria to be a case of hypothyroidism were identified.
Arm/Group | Hypothyroidism Cases With CT Scan | Hypothyroidism Cases With Cardiac Catheterization
Number analyzed (Participants) | 18 | 16
Participants
  <30 days | 4 | 3
  30 - 59 days | 4 | 3
  60+ days | 10 | 10

8. Secondary Outcome: Classification of Subclinical/Manifest Hypothyroidism by Type of Exposure
Time Frame: Up to 365 days after a diagnostic scan with iodinated contrast agent
Measure: Count of Participants; unit: Participants
Arm/Group | Hypothyroidism Cases With CT Scan | Hypothyroidism Cases With Cardiac Catheterization
Number analyzed (Participants) | 18 | 16
Participants
  Subclinical hypothyroidism | 15 | 9
  Manifest hypothyroidism | 2 | 1
  Treatment or diagnosis with no TSH test | 1 | 6

9. Secondary Outcome: Classification of Hypothyroidism by Etiology
Time Frame: Up to 365 days after a diagnostic scan with iodinated contrast agent
Measure: Count of Participants; unit: Participants
Arm/Group | Hypothyroidism Cases
Number analyzed (Participants) | 34
Participants
  Iodine induced cases | 23
  Other etiology cases | 11

ADVERSE EVENTS:
Time Frame: Incidence of hypothyroidism was assessed up to one year after iodine contrast exposure
Description: This study is a retrospective study using data from the database in United States. The safety outcome focused on the incidence of hypothyroidism for up to one year after iodine contrast exposure. Please refer to the result of primary outcome measure. All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed during this retrospective observation study. Only retrospective safety outcome data were assessed, which are on the outcome measures module.
Arm/Group | Iodine Contrast Agent
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-11): https://cdn.clinicaltrials.gov/large-docs/27/NCT02959827/Prot_SAP_000.pdf